CLINICAL TRIAL: NCT05369988
Title: VALIDATION OF THE VIBe INTRAOPERATIVE BLEEDING SCALE IN LIVER SURGERY. PROSPECTIVE AND MULTICENTRIC STUDY
Brief Title: VALIDATION OF THE VIBe INTRAOPERATIVE BLEEDING SCALE IN LIVER SURGERY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other)
Responsible Party: Principal Investigator, Mario Serradilla, MD, FACS, MD, FACS, Hospital Miguel Servet
Other Study IDs: PI21-510
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Surgical Hemorrhage; Liver Cancer; Liver Metastases
Keywords: Liver surgery; Surgical hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical hemostasis has become one of the fundamental principles for the advancement of surgery. The use of hemostatic agents is standard in many surgical specialties, although the lack of consensus or standardized classifications to determine intraoperative bleeding has led to their inappropriate selection on many occasions. The recommendations of international organizations highlight the need for a bleeding severity scale validated in clinical studies that allows selecting the hemostatic agent that best suits each case.

DETAILED DESCRIPTION:
Surgical hemostasis has become one of the fundamental principles for the advancement of surgery. The use of hemostatic agents is standard in many surgical specialties, with greater use in major surgeries. Inadequate hemostasis significantly increases the risk of perioperative morbidity and mortality, healthcare costs and the use of resources. The need for hemostasis has led to the development of various topical hemostatic agents.

Clinical studies that have analyzed the use of topical hemostats have not used standardized definitions or classifications to determine the severity of intraoperative bleeding, partly due to a lack of consensus on the definition of the severity of bleeding and partly due to the severity of bleeding. lack of requirements to do so. This has led many surgeons to an inadequate selection of hemostats for different bleeding situations, the results being inefficient. Using standardized criteria, the results of clinical studies can be compared to determine the effectiveness of hemostatic agents.

The FDA (Food and Drug Administration) requires the use of a bleeding severity scale validated in clinical studies investigating hemostatic agents. The VIBe (Validated Intraoperative Bleeding Scale) for intraoperative bleeding was developed in 2017.This scale has been validated by a large number of expert surgeons from all specialties, but in an animal model. However, it has not yet been clinically validated.

Liver surgery is one of the surgeries where intraoperative bleeding is more important. In Spain, around 5000 liver resections are performed annually, not including liver transplants. It is, therefore, a perfect framework to validate the applicability of the VIBe scale of severity of intraoperative bleeding.

In order to evaluate the viability of a prospective clinical study in liver surgery, a parallel project has been worked on based on the evaluation of the applicability of the VIBe scale, carried out by liver surgeons by reviewing the original video recordings described in the VIBe scale. Forty-seven surgeons were selected from 10 medium-high-volume liver surgery centers, all of them reference centers (same centers that will participate in the prospective study). 5 of the 10 hospitals perform liver transplants. These centers have a mean reference population of 922,506 ± 225,603 patients. The mean number of major hepatectomies per year is 23 ± 16, the number of minor hepatectomies 56 ± 24, and the number of liver transplants 40 ± 27. 40.5% of all hepatectomies are performed by a minimally invasive approach.

The 47 surgeons viewed 14 videos used by Lewis et al. for the validation of the original VIBe scale. 63.3% of the participating surgeons were men with a mean age of 41.6 years. 17% were unit / department heads and 83% were senior surgeons. The mean experience was 9.3 years, and the majority were experts (21.3%) or with advanced knowledge (53.2%) in minimally invasive surgery. Only 23.4% had prior knowledge of the VIBe scale, but all surgeons used hemostats in their daily clinical practice. The VIBe scale achieved a mean intraobserver agreement of 0.985 and an interobserver agreement of 0.929, neither of which was influenced by the experience of the surgeon or the volume of surgeries per year. The average rating for all videos was 67% correct, in line with the original validation. Most surgeons considered that the scale represented the range of severity of bleeding in their procedures (91%), relevant to assess intraoperative hemostasis in clinical studies (96%) and clinical practice (87.2%), useful in CMI (96%), and also to differentiate hemostatic agents (81%).

With these preliminary data, based on the video classification exercise, we can conclude that the VIBe scale is useful for the assessment of the severity of bleeding performed by liver surgeons. Therefore, an assessment of the severity of intraoperative bleeding using the scale in actual liver surgery is feasible. Our goal is to publish these results independently before starting the clinical observation record.

To evaluate the clinical applicability, a prospective registry of patients undergoing liver surgery has been designed in the 10 selected Spanish centers. Demographic and preoperative, intraoperative and postoperative data will be collected. Intraoperative bleeding will be measured according to the VIBe scale at two points of the surgical intervention: the maximum bleeding and at the end of the surgery. Data will be collected on the type of hemostatic or surgical strategy that has been carried out to correct bleeding (i.e. pressure, suture, coagulation, hemostatic, etc.) and other data related to bleeding (blood loss, units of blood transfused, etc.). Postoperative complications will be classified according to the Clavien-Dindo classification and the CCI (Comprehensive Complication Index). Major complications are defined as those with a Clavien-Dindo ≥ IIIa. The classification of liver failure and postoperative bleeding are defined following the International Study Group of Liver Liver Surgery (ISGLS) classifications. At the end of the registration a statistical analysis of the data will be performed to determine the applicability and usefulness of the VIBe scale in liver surgery, as well as to determine the relationship between the type of bleeding, the hemostatic measurements used, the success rate of the hemostatic measurements, and the bleeding-related complications.

Despite the extensive literature published on liver surgery, there is no scientific evidence that allows us to have validated scalds that quantify the severity of intraoperative bleeding and, consequently, select which is the best hemostatic procedure that is adapted to each case. All of this has repercussions on patient safety, increased postoperative morbidity and mortality, as well as the inappropriate use of healthcare resources and consequently increased costs.

This prospective multicenter study in national centers that perform Liver Surgery aims to evaluate and validate a scale that allows quantifying intraoperative bleeding in liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18, scheduled for liver surgery, by open or minimally invasive approach, regardless of diagnosis;
* ASA score <4
* They have signed the informed consent.

Exclusion Criteria:

* Patients with contraindications for liver surgery
* Emergency surgical interventions
* Patients <18 years
* Patients who have not signed the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry includes all the elderly patients operated on in the participating Spanish centers who underwent liver surgery in the period described and that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
To validate the VIBe scale. | 30 days
  To validate the VIBe scale for intraoperative bleeding in liver surgery.

SECONDARY OUTCOMES:
Usefulness of the scale | 30 days
  Assess the repeatability, reproducibility and usefulness of the scale in this type of surgery.
Determine the relationship between type of bleeding and hemostatic used, the success rate of hemostatic measurements, and complications related to bleeding. | 30 days
  Determine the relationship between type of bleeding and hemostatic used, the success rate of hemostatic measurements, and complications related to bleeding.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Mario Serradilla Martin, Zaragoza
  - Daniel Aparicio Lopez, Zaragoza

REFERENCES:
- [Result] American Society of Anesthesiologists Task Force on Perioperative Blood Management. Practice guidelines for perioperative blood management: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Management*. Anesthesiology. 2015 Feb;122(2):241-75. doi: 10.1097/ALN.0000000000000463. No abstract available. PMID 25545654
- [Result] Wright Jr. JR, Schachar, NS. Necessity is the mother of invention: William Stewart Halsted's addiction and its influence on the development of residency training in North America. Can J Surg. 2020 Jan 16;63(1):E13-E19. doi: 10.1503/cjs.003319. PMID 31944636
- [Result] Shander A, Van Aken H, Colomina MJ, Gombotz H, Hofmann A, Krauspe R, Lasocki S, Richards T, Slappendel R, Spahn DR. Patient blood management in Europe. Br J Anaesth. 2012 Jul;109(1):55-68. doi: 10.1093/bja/aes139. Epub 2012 May 24. PMID 22628393
- [Result] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Brown JR, Despotis GJ, Hammon JW, Reece TB, Saha SP, Song HK, Clough ER; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Shore-Lesserson LJ, Goodnough LT, Mazer CD, Shander A, Stafford-Smith M, Waters J; International Consortium for Evidence Based Perfusion; Baker RA, Dickinson TA, FitzGerald DJ, Likosky DS, Shann KG. 2011 update to the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesiologists blood conservation clinical practice guidelines. Ann Thorac Surg. 2011 Mar;91(3):944-82. doi: 10.1016/j.athoracsur.2010.11.078. PMID 21353044
- [Result] Menkis AH, Martin J, Cheng DC, Fitzgerald DC, Freedman JJ, Gao C, Koster A, Mackenzie GS, Murphy GJ, Spiess B, Ad N. Drug, devices, technologies, and techniques for blood management in minimally invasive and conventional cardiothoracic surgery: a consensus statement from the International Society for Minimally Invasive Cardiothoracic Surgery (ISMICS) 2011. Innovations (Phila). 2012 Jul-Aug;7(4):229-41. doi: 10.1097/IMI.0b013e3182747699. PMID 23123988
- [Result] Kommu SS, McArthur R, Emara AM, Reddy UD, Anderson CJ, Barber NJ, Persad RA, Eden CG. Current Status of Hemostatic Agents and Sealants in Urologic Surgical Practice. Rev Urol. 2015;17(3):150-9. PMID 26543429
- [Result] Wright JD, Ananth CV, Lewin SN, Burke WM, Siddiq Z, Neugut AI, Herzog TJ, Hershman DL. Patterns of use of hemostatic agents in patients undergoing major surgery. J Surg Res. 2014 Jan;186(1):458-66. doi: 10.1016/j.jss.2013.07.042. Epub 2013 Aug 13. PMID 23993203
- [Result] Dimick JB, Chen SL, Taheri PA, Henderson WG, Khuri SF, Campbell DA Jr. Hospital costs associated with surgical complications: a report from the private-sector National Surgical Quality Improvement Program. J Am Coll Surg. 2004 Oct;199(4):531-7. doi: 10.1016/j.jamcollsurg.2004.05.276. PMID 15454134
- [Result] Shander A. Financial and clinical outcomes associated with surgical bleeding complications. Surgery. 2007 Oct;142(4 Suppl):S20-5. doi: 10.1016/j.surg.2007.06.025. PMID 18019945
- [Result] Christensen MC, Krapf S, Kempel A, von Heymann C. Costs of excessive postoperative hemorrhage in cardiac surgery. J Thorac Cardiovasc Surg. 2009 Sep;138(3):687-93. doi: 10.1016/j.jtcvs.2009.02.021. Epub 2009 Apr 19. PMID 19698857
- [Result] Stokes ME, Ye X, Shah M, Mercaldi K, Reynolds MW, Rupnow MF, Hammond J. Impact of bleeding-related complications and/or blood product transfusions on hospital costs in inpatient surgical patients. BMC Health Serv Res. 2011 May 31;11:135. doi: 10.1186/1472-6963-11-135. PMID 21627788
- [Result] Levy JH, Dutton RP, Hemphill JC 3rd, Shander A, Cooper D, Paidas MJ, Kessler CM, Holcomb JB, Lawson JH; Hemostasis Summit Participants. Multidisciplinary approach to the challenge of hemostasis. Anesth Analg. 2010 Feb 1;110(2):354-64. doi: 10.1213/ANE.0b013e3181c84ba5. Epub 2009 Dec 10. PMID 20007735
- [Result] Filipescu DC, Stefan MG, Valeanu L, Popescu WM. Perioperative management of antiplatelet therapy in noncardiac surgery. Curr Opin Anaesthesiol. 2020 Jun;33(3):454-462. doi: 10.1097/ACO.0000000000000875. PMID 32371645
- [Result] Schuhmacher C, Pratschke J, Weiss S, Schneeberger S, Mihaljevic AL, Schirren R, Winkler M, Emmanouilidis N. Safety and effectiveness of a synthetic hemostatic patch for intraoperative soft tissue bleeding. Med Devices (Auckl). 2015 Mar 31;8:167-74. doi: 10.2147/MDER.S79556. eCollection 2015. PMID 25878513
- [Result] Fischer CP, Bochicchio G, Shen J, Patel B, Batiller J, Hart JC. A prospective, randomized, controlled trial of the efficacy and safety of fibrin pad as an adjunct to control soft tissue bleeding during abdominal, retroperitoneal, pelvic, and thoracic surgery. J Am Coll Surg. 2013 Sep;217(3):385-93. doi: 10.1016/j.jamcollsurg.2013.02.036. PMID 23969113
- [Result] Lewis KM, Li Q, Jones DS, Corrales JD, Du H, Spiess PE, Lo Menzo E, DeAnda A Jr. Development and validation of an intraoperative bleeding severity scale for use in clinical studies of hemostatic agents. Surgery. 2017 Mar;161(3):771-781. doi: 10.1016/j.surg.2016.09.022. Epub 2016 Nov 10. PMID 27839931
- [Derived] Aparicio-Lopez D, Asencio-Pascual JM, Blanco-Fernandez G, Cugat-Andorra E, Gomez-Bravo MA, Lopez-Ben S, Martin-Perez E, Sabater L, Ramia JM, Serradilla-Martin M. Evaluation of the validated intraoperative bleeding scale in liver surgery: study protocol for a multicenter prospective study. Front Surg. 2023 Oct 2;10:1223225. doi: 10.3389/fsurg.2023.1223225. eCollection 2023. PMID 37850041

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT05369988/Prot_SAP_ICF_000.pdf